CLINICAL TRIAL: NCT07115901
Title: Guaranteed Income to Boost HIV Care Continuity and Suppression Post-Jail Release
Acronym: GI-BOOST
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 25-43573; H25EJ9047 (Other Grant/Funding Number: California HIV/AIDS Research Program)
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: HIV (Human Immunodeficiency Virus)
Keywords: HIV; Guaranteed Income; Criminal Legal Involvement
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lump sum (Experimental): Participants receive the full guaranteed income amount ($6,750) as one lump sum payment at the beginning of the study.
  Interventions: Other: Guaranteed Income
- Monthly Installments (Experimental): Participants receive the guaranteed income intervention split into 9-monthly installments of $750/month
  Interventions: Other: Guaranteed Income
- Choice (Experimental): Participants choose which method of Guaranteed Income disbursement they will receive (either lump sum or monthly installments).
  Interventions: Other: Guaranteed Income

INTERVENTIONS:
Other: Guaranteed Income — Participants will receive guaranteed income (GI) to the amount of $6,750 over the study period. While all participants will receive the GI intervention, there will be variation in the method of disbursement. Some participants will receive the GI as a one-time lump sum payment whereas other participants will receive the same GI amount split into 9-monthly installments.

SUMMARY:
The goal of this clinical trial is to understand the implementation requirements and potential health impacts of a guaranteed income (GI) intervention targeting people living with HIV with criminal legal involvement (PWH-CLI). The main questions it aims to answer are:

* How acceptable is a GI intervention, and its intervention components, among PWH-CLI participants and stakeholders?
* How feasible is a GI intervention for PWH-CLI? What are the implementation barriers and opportunities for this intervention?
* What is the preliminary efficacy of the GI intervention on improving HIV care outcomes for PWH-CLI? Researches will compare study engagement and study outcomes across three randomization arms (A: receive full GI amount as one lump sum payment; B: receive full GI amount split over nine monthly installments; C: participant chooses whether to receive GI as lump sum payment or monthly installments). HIV care outcomes will be compared against a retrospective cohort of PWH-CLI patients as historical controls.

Participants will:

* Be randomized to receive GI intervention as a lump sum payment or monthly installment (over nine months) or choose their preference.
* Complete 3 surveys throughout study follow up to assess experience with the intervention, experience with social services and benefits programs, experience with the criminal legal system, and HIV care outcomes.
* Be interviewed by the research team to further understand the experience with the intervention.

DETAILED DESCRIPTION:
One-in-seven people living with HIV (PWH) experience incarceration annually. HIV prevalence among those with criminal legal involvement (CLI) is 3x higher than the general population. Upon release, PWH-CLI encounter competing priorities and structural barriers to addressing unmet basic needs, resulting in suboptimal care cascade outcomes. Guaranteed income (GI) through unconditional cash transfers can improve mental health, meet basic needs, and boost employment prospects. However, its effects on PWH-CLI, who face unique post-release challenges affecting HIV treatment retention and viral suppression, remain uncharacterized.

Our three-arm pilot study will assess the feasibility, acceptability, implementation requirements, and preliminary efficacy of a GI intervention to improve HIV care in PWH-CLI released from the San Francisco County (SFC) jail. We will randomize up to 39 very low-income patients discharged to a SFDPH network HIV clinic to 1 of 3 arms: A) one lump-sum payment of $6,750; B) 9-monthly installments of $750; or C) "preference" (patient chooses either A or B). We will offer opt-in financial mentoring (FM) sessions during the pilot to bolster GI impacts. Clinical appointment and viral load outcome data will be collected from medical records. All patients will complete quantitative surveys (1 baseline, 2 follow-up) to assess GI experience, patient context, and acceptability. Baseline and endline qualitative interviews with patients (n=12; 4/arm) will explore the GI experience, impacts on HIV treatment, and critical implementation questions to inform future research and policy. Qualitative interviews with system partners (n=10) will explore community perceptions of GI and opportunities to integrate GI in HIV programming and policy.

Given PWH-CLI's economic and social marginalization, we will leverage our existing retrospective cohort of PWH-CLI released from SFC jail as historical controls to test preliminary efficacy against pilot participants - comparing clinical appointments and viral load - instead of utilizing a concurrent no-GI control group. Variation in GI disbursement will provide needed data on acceptability and preliminary efficacy of distribution modes and the role of patient agency in pilot outcomes and overall engagement.

We will pilot a GI intervention for PWH-CLI leaving SFC jail, aiming to reduce structural barriers to care and improve HIV care cascade engagement. Our specific aims are to:

(Aim 1) Determine GI intervention acceptability among PWH-CLI and stakeholders. We will explore patient preference for GI disbursement and if GI mode impacts successful HIV care engagement and study procedures through longitudinal qualitative interviews. Thematic analysis will elucidate individual impacts of GI amidst contextual facilitators and barriers to care. Qualitative interviews with system partners will gauge community and policy perceptions of GI intervention acceptability and optimal means to integrate.

(Aim 2) Assess GI intervention feasibility and implementation barriers/opportunities for PWH-CLI. Feasibility measures include differences in study engagement (FM uptake, surveys) by randomization arm. We will assess reported GI receipt experience for PWH-CLI who do/not access other safety net programs and for those experiencing unstable housing, residential treatment programs, and re-incarceration to understand overlap and benefit combinations with other state/county programs to optimize future implementation.

(Aim 3) Test preliminary efficacy of the GI intervention on improving HIV care outcomes. By randomization arm, we will compare the percentage linked to an HIV care provider within 30 days of jail release, retained in HIV care (>= 2 visit >=90 days apart), and virally suppressed at 9 months. GI pilot HIV cascade outcomes will be compared to propensity-matched historical controls from our retrospective cohort of PWH-CLI. We will also assess group differences in re-incarceration rates.

A significant subset of PWH, PWH-CLI are among the least retained in HIV care and adherent to ART. This research will bridge current knowledge gaps by testing GI implementation strategies, assessing community support and integration opportunities, and testing preliminary efficacy in HIV care outcomes to inform a large-scale trial.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for this pilot study if they are 18 years of age or older, are living with an HIV diagnosis, have a recent incarceration in the San Francisco County Jail (within three months of study enrollment), and qualify as very low income (for example, currently experiencing homelessness or having an income less than 30% of the area median income). Participants must be English literate.

Exclusion Criteria:

* Individuals with an active psychosis who are not on treatment will be ineligible to enroll in the study (however, individuals with a psychiatric co-morbidity who are on treatment will remain eligible). For the purpose of the Focus Care enrollment (the method of GI disbursement), individuals who do not have a social security number or individual tax ID number will be ineligible for this pilot study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
HIV viral suppression | From enrollment to end of the intervention at 9 months
  Percent of participants (total and by randomization arm) that are HIV virally suppressed at 9 months

SECONDARY OUTCOMES:
Linkage to HIV care | From enrollment to one month after enrollment
  Percentage of participants (in total and by randomization arm) that have linked to an HIV care provider within one month of study enrollment
Retention in HIV care | From enrollment to end of intervention at 9 months
  Percent of participants (in total and by randomization arm) that are retained in HIV care (defined as two or more HIV care visits and/or viral load measurements at least 90 days apart from each other) at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Wesson, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Given the small projected sample size for this pilot study (n=33) and the vulnerable nature of the study population (people living with HIV with recent criminal legal involvement), we do not have plans to share IPD in order to protect participant anonymity.

REFERENCES:
- [Background] Delevry D, Le QA. Effect of Treatment Preference in Randomized Controlled Trials: Systematic Review of the Literature and Meta-Analysis. Patient. 2019 Dec;12(6):593-609. doi: 10.1007/s40271-019-00379-6. PMID 31372909
- [Background] West S, Castro A. Impact of Guaranteed Income on Health, Finances, and Agency: Findings from the Stockton Randomized Controlled Trial. J Urban Health. 2023 Apr;100(2):227-244. doi: 10.1007/s11524-023-00723-0. Epub 2023 Apr 10. PMID 37037977
- [Background] Moher M, Erickson M, Black P, Price M, Fraser C, Norman WV, Guillemi S, Pick N, Elwood Martin R. Improving Post-Release Care Engagement for People Living with HIV Involved in the Criminal Justice System: A Systematic Review. AIDS Behav. 2022 May;26(5):1607-1617. doi: 10.1007/s10461-021-03513-4. Epub 2021 Oct 27. PMID 34705154
- [Background] Iroh PA, Mayo H, Nijhawan AE. The HIV Care Cascade Before, During, and After Incarceration: A Systematic Review and Data Synthesis. Am J Public Health. 2015 Jul;105(7):e5-16. doi: 10.2105/AJPH.2015.302635. Epub 2015 May 14. PMID 25973818
- [Background] Badowski ME, Patel M. Evaluation of Immunologic and Virologic Function in Reincarcerated Patients Living With HIV or AIDS. J Correct Health Care. 2022 Jun;28(3):203-206. doi: 10.1089/jchc.20.07.0055. Epub 2022 Apr 21. PMID 35447035